CLINICAL TRIAL: NCT03329352
Title: Evaluation of a Full-Face Mask for the Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-227
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2021-09-21 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: After a period of baseline, all enrolled participants will be put on the same trial mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- F&P Full-Face Mask (Experimental): Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial full-face mask during this treatment arm. Participants on the extension will use for a further six months after Visit 3.
  Interventions: Device: F&P Full-Face Mask

INTERVENTIONS:
Device: F&P Full-Face Mask — The F&P full-face mask will serve as the participant's primary PAP therapy mask for the duration of the trial period (from Visit 2 to Visit 3). For participants taking part in the study extension, they will be using the trial full-face mask as their primary PAP therapy mask for 6 months after Visit 3.

SUMMARY:
The investigation is designed to evaluate the comfort, ease of use and performance of a trial nasal mask for the treatment of Obstructive Sleep Apnea (OSA) in the home environment.

DETAILED DESCRIPTION:
The investigation is a prospective, non-randomized, non-blinded study. Up to 45 OSA participants who currently use a full-face mask will be recruited.

The study will involve a baseline (Visit 1) data gathering with the participant's PAP therapy and their usual mask. This will be followed by the participants being fitted with the trial full-face mask by a sleep technician for use in-home (Visit 2). The participant then will come in to return the mask (Visit 3) and give feedback on their experience using the mask in home in the form of a structured interview during Visit 3. If the participants prefer the trial full-face mask they will be asked if they would like to continue using the trial mask for a further six months in home. There will be a follow up phone call gain feedback or address any issues at months 2 and 4 of the six month extension period. At the end of the six month extension period, the participants will return the trial full-face mask to NTLSC and answer a few questions around their feedback on the mask after using it for six months.

The mask and CPAP (if used from the loan research pool) will be returned to the institution at the conclusion of the trial and participant will return to their usual mask and therapy device for the treatment of Obstructive Sleep Apnea.

Neither the investigators nor the participants will be blinded to the study.

Data from initial 2 week trial is reported here.

ELIGIBILITY:
Inclusion Criteria:

* AHI ≥ 5 from diagnostic PSG night
* Aged 22 and over (FDA defined as adult)
* Either prescribed APAP, CPAP or Bi-Level PAP for OSA
* Existing full-face mask users
* Fluent in spoken and written English

Exclusion Criteria:

* Inability to give informed consent
* Patient intolerant to CPAP therapy
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or CO2 retention
* Pregnant or think they may be pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ostransky, MD, Principal Investigator — Board Certified Sleep Specialist
Locations (1):
- North Texas Lung and Sleep Clinic, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with any other researchers or organizations.

RESULTS

PARTICIPANT FLOW:
Groups:
- F&P Toffee Full-Face Mask: Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial full-face mask during this treatment arm. Participants on the extension will use for a further six months after Visit 3.
  F&P Toffee Full-Face Mask: The F&P Toffee full-face mask will serve as the participant's primary PAP therapy mask for the duration of the trial period (from Visit 2 to Visit 3).
Period: F&P Toffee Full Face Mask Validation
Arm/Group | F&P Toffee Full-Face Mask
Started | 44
Completed | 42
Not Completed | 2
Period: Extension
Arm/Group | F&P Toffee Full-Face Mask
Started | 29
Completed | 22
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- F&P Toffee Full-Face Mask: Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial full-face mask during this treatment arm. Participants on the extension will use for a further six months after Visit 3.
  F&P Toffee Full-Face Mask: The F&P Toffee Full-face mask will serve as the participant's primary PAP therapy mask for the duration of the trial period (from Visit 2 to Visit 3). For participants taking part in the study extension, they will be using the trial full-face mask as their primary PAP therapy mask for 6 months after Visit 3.
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Trial Mask Comfort
Description: Determined from questionnaire - Subjective Uses a 5 point Likert Scale (Very Uncomfortable, Uncomfortable, Same as usual, Comfortable, Very Comfortable).
Time Frame: 14 ± 5 days in-home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 42
Participants
  Very comfortable | 20
  Comfortable | 16
  Neutral | 4
  Uncomfortable | 1
  Very uncomfortable | 0
  N/A | 1

2. Primary Outcome: Participant Count of Acceptable Trial Mask Performance - Objective
Description: Determined from AHI data, a measure of disease severity, recorded from the PAP device - Objective
Time Frame: 14 ± 5 days in-home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 42
Participants
  Pass | 34
  Fail | 0
  N/A | 8

3. Primary Outcome: Trial Mask Seal Performance - Subjective
Description: Determined from questionnaire - Subjective Uses a 5 point Likert Scale
Time Frame: 14 ± 5 days in-home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 42
Participants
  Very good | 17
  Good | 14
  Neutral | 4
  Poor | 4
  Very poor | 2
  N/A | 1

4. Primary Outcome: Trial Mask Ease of Cleaning
Description: Determined from questionnaires - Subjective
  A single question asked participants to report their ability to clean the mask on a 5 point Likert Scale with scores ranging from very easy, easy, neutral, hard, and very hard.
Time Frame: 14 ± 5 days in-home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 42
Participants
  Very easy | 25
  Easy | 15
  Neutral | 2
  Hard | 0
  Very hard | 0

5. Primary Outcome: Trial Mask Ease-of-use
Description: Participants experience removing mask from face, determined from questionnaires and a sleep diary - Subjective Uses a 5 point Likert Scale. Also includes, discussion questions around comfort.
Time Frame: 14 ± 5 days in-home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 42
Participants
  Very easy | 27
  Easy | 14
  Neutral | 1
  Hard | 0
  Very hard | 0

6. Secondary Outcome: Participant Count of Acceptable Mask Leak
Description: Data recorded from PAP device reporting amount of air leaking from the mask during PAP therapy. If mask leak was over 60 L/min it was compared to the participants baseline leak values to assess if mask leak with the trial mask was acceptable or not.
Time Frame: 14 ± 5 days in-home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 42
Participants
  Pass | 30
  Fail | 4
  N/A | 8

7. Secondary Outcome: Participant Count of Seal Size Determination
Description: Whether the sizing guide prediction tool used to size participants matched the trial administrators sizing prediction.
Time Frame: 1 day-time appointment (1 hour) Visit 2
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Full-Face Mask
Number analyzed (Participants) | 44
Participants
  Pass | 28
  Fail | 16

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 6 months the trial ran for (including the extension)
Groups:
- F&P Full-Face Mask: Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial full-face mask during this treatment arm. Participants on the extension will use for a further six months after Visit 3.
  F&P Full-Face Mask: The F&P full-face mask will serve as the participant's primary PAP therapy mask for the duration of the trial period (from Visit 2 to Visit 3). For participants taking part in the study extension, they will be using the trial full-face mask as their primary PAP therapy mask for 6 months after Visit 3.
  Adverse event data will be collated for both arms of the trial for simplicity.
Arm/Group | F&P Full-Face Mask
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 2/42
Other Adverse Events (participants affected / at risk) | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F&P Full-Face Mask (N=42)
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1) — Admitted to ER, was note related to the trial and resolved no sequel
Myocardial infarction (Cardiac disorders) | 1 (1) — Admitted to ICU. Not related to trial and resolved no sequel
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F&P Full-Face Mask (N=42)
Facial irritation (Skin and subcutaneous tissue disorders) | 2 (2) — Irritations were present whilst using their usual mask so reported as not related and resolved no sequel

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03329352/Prot_000.pdf